CLINICAL TRIAL: NCT01210456
Title: The Prevention Contrast-Induced Acute Kidney Injury With the Triple Combination of Hydration With Physiological Saline, N-Acetylcysteine and Sodium Bicarbonate
Brief Title: Efficacy Trial of N-Acetylcysteine and Sodium Bicarbonate for the Prevention of Contrast-Induced Acute Kidney Injury
Acronym: PREKIT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tokushukai Medical Group (Other)
Responsible Party: Principal Investigator, Daisuke Hachinohe, Sapporo Higashi Tokushukai Hospital, Tokushukai Medical Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREKIT-001
Record Dates: First submitted 2010-07-11; First posted 2010-09-28 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Contrast Media; Acute Kidney Injury; N-Acetylcysteine; Bicarbonate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury | interventions — Acetylcysteine; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiological Saline and N-Acetylcysteine (Active Comparator)
  Interventions: Drug: Physiological Saline, N-Acetylcysteine and Sodium Bicarbonate
- Physiological Saline, N-Acetylcysteine and Sodium Bicarbonate (Active Comparator)
  Interventions: Drug: Physiological Saline, N-Acetylcysteine and Sodium Bicarbonate

INTERVENTIONS:
Drug: Physiological Saline, N-Acetylcysteine and Sodium Bicarbonate — All patients receive N-Acetylcysteine(NAC) and sodium chloride. NAC is given orally at a dose of 700mg twice daily, on the day before and on the day of administration of the contrast media, for a total of two days.
  154mEq/L of sodium chloride is given intravenously. The initial intravenous bolus is 3ml/kg per hour for 1 hour immediately before contrast injection. And then, patients receive the same fluid at 1ml/kg per hour during the contrast exposure and for 6 hours after the procedure.
  In addition, intervention arms receive sodium bicarbonate.1000mEq/L of sodium bicarbonate is given intravenously twice at a dose of 40ml immediately before the contrast exposure and immediately after the procedure.

SUMMARY:
Contrast-Induced Acute Kidney Injury(CIAKI) was defined as an absolute increase in serum creatinine of more than or equal to 0.3mg/dl (≥ 26.4 μmol/l), a percentage increase in serum creatinine of more than or equal to 50% (1.5-fold from baseline) within 48 hours of intravascular contrast administration in the absence of any alternative causes, or a reduction in urine output documented oliguria of less than 0.5 ml/kg per hour for more than six hours.

It is the common cause of new hospital-acquired renal insufficiency. The occurrence of CIAKI may be influenced by pre-existing renal insufficiency, diabetic nephropathy, dehydration, congestive heart failure, concurrent administration of nephrotoxic drugs, or the dose and type of contrast media used. Previous studies have shown the independent effectiveness of several agents in preventing CIAKI.

Even now, hydration is crucial for preventing CIAKI. Since CIAKI is presumed to be caused by free radical generation, N-Acetylcysteine, which is a potent free radical scavenger, is shown to be effective in preventing nephropathy. At the same time, because free radical formation is promoted by an acidic environment, bicarbonate, which alkalinizes renal tubular fluid, has been shown to reduce renal involvement.

These days, some studies have shown that hydration with sodium bicarbonate plus N-Acetylcysteine was effective and safe in the prevention of CIAKI. In these studies, bicarbonate was used for both alkalinizing renal tubular fluid and hydration. However, if we want to do hydration, we can use saline and if we want to alkalinize renal tubular fluid, we might use bicarbonate by bolus injection.

Actually, bicarbonate for hydration is prepared at sterile preparation room in a hospital, which is very cumbersome procedure and increase in cost. This is one of the reasons that bicarbonate for hydration use does not become common with wide clinical application.

In past issues, though it differs depending on the level of the renal dysfunction, the probability of CIAKI was 8-33% when hydration was administered, 5-15% when hydration and N-Acetylcysteine were administered, and 1.8-1.9% when bicarbonate and N-Acetylcysteine were administered.

Thus, we can hypothesize the combination of N-Acetylcysteine and bicarbonate will play a complementary role in preventing contrast-induced nephropathy.

This is the rational for this study.

ELIGIBILITY:
Inclusion Criteria:

* serum creatinine more or equal than 1.1mg/dL
* procedures using contrast media

Exclusion Criteria:

* congestive heart failure
* serum creatinine less than 1.1mg/dl
* allergy to contrast media
* preexisting dialysis
* emergency catheterization
* recent exposure to contrast within 2 days of the study
* refuse to entry this study
* PTRA
* dialysis after procedure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2009-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Development of contrast-induced acute kidney injury | within 48 hours
  Contrast-Induced Acute Kidney Injury(CIAKI) was defined as an absolute increase in serum creatinine of more than or equal to 0.3mg/dl (≥ 26.4 μmol/l), a percentage increase in serum creatinine of more than or equal to 50% (1.5-fold from baseline) within 48 hours of intravascular contrast administration in the absence of any alternative causes, or a reduction in urine output documented oliguria of less than 0.5 ml/kg per hour for more than six hours.

SECONDARY OUTCOMES:
Requirement of dialysis | 6 months
Requirement of hospitalization and death | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daisuke Hachinohe, MD, Principal Investigator — Sapporo Higashi Tokushukai Hospital
Locations (1):
- Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido, Japan

REFERENCES:
- [Background] Morcos SK. Contrast media-induced nephrotoxicity--questions and answers. Br J Radiol. 1998 Apr;71(844):357-65. doi: 10.1259/bjr.71.844.9659127.
- [Background] Benko A, Fraser-Hill M, Magner P, Capusten B, Barrett B, Myers A, Owen RJ; Canadian Association of Radiologists. Canadian Association of Radiologists: consensus guidelines for the prevention of contrast-induced nephropathy. Can Assoc Radiol J. 2007 Apr;58(2):79-87. PMID 17521052
- [Background] Hou SH, Bushinsky DA, Wish JB, Cohen JJ, Harrington JT. Hospital-acquired renal insufficiency: a prospective study. Am J Med. 1983 Feb;74(2):243-8. doi: 10.1016/0002-9343(83)90618-6. PMID 6824004
- [Background] Morcos SK, Thomsen HS, Webb JA. Contrast-media-induced nephrotoxicity: a consensus report. Contrast Media Safety Committee, European Society of Urogenital Radiology (ESUR). Eur Radiol. 1999;9(8):1602-13. doi: 10.1007/s003300050894. PMID 10525875
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Background] Briguori C, Tavano D, Colombo A. Contrast agent--associated nephrotoxicity. Prog Cardiovasc Dis. 2003 May-Jun;45(6):493-503. doi: 10.1053/pcad.2003.YPCAD16. PMID 12800130
- [Background] Rihal CS, Textor SC, Grill DE, Berger PB, Ting HH, Best PJ, Singh M, Bell MR, Barsness GW, Mathew V, Garratt KN, Holmes DR Jr. Incidence and prognostic importance of acute renal failure after percutaneous coronary intervention. Circulation. 2002 May 14;105(19):2259-64. doi: 10.1161/01.cir.0000016043.87291.33. PMID 12010907
- [Background] Iakovou I, Dangas G, Mehran R, Lansky AJ, Ashby DT, Fahy M, Mintz GS, Kent KM, Pichard AD, Satler LF, Stone GW, Leon MB. Impact of gender on the incidence and outcome of contrast-induced nephropathy after percutaneous coronary intervention. J Invasive Cardiol. 2003 Jan;15(1):18-22. PMID 12499523
- [Background] Marenzi G, Assanelli E, Marana I, Lauri G, Campodonico J, Grazi M, De Metrio M, Galli S, Fabbiocchi F, Montorsi P, Veglia F, Bartorelli AL. N-acetylcysteine and contrast-induced nephropathy in primary angioplasty. N Engl J Med. 2006 Jun 29;354(26):2773-82. doi: 10.1056/NEJMoa054209. PMID 16807414
- [Background] Detrenis S, Meschi M, Musini S, Savazzi G. Lights and shadows on the pathogenesis of contrast-induced nephropathy: state of the art. Nephrol Dial Transplant. 2005 Aug;20(8):1542-50. doi: 10.1093/ndt/gfh868. No abstract available. PMID 16033768
- [Background] Goss RJ. Photoperiodic control of antler cycles in deer. III. Decreasing versus increasing day lengths. J Exp Zool. 1976 Sep;197(3):307-12. doi: 10.1002/jez.1401970302. PMID 965912
- [Background] Nazarko L. Working parents: a woman's rightful place. Nurs Stand. 1992 May 6-12;6(33):46. doi: 10.7748/ns.6.33.46.s39. No abstract available. PMID 1591186
- [Background] Itoh Y, Yano T, Sendo T, Oishi R. Clinical and experimental evidence for prevention of acute renal failure induced by radiographic contrast media. J Pharmacol Sci. 2005 Apr;97(4):473-88. doi: 10.1254/jphs.crj05002x. Epub 2005 Apr 9. PMID 15821342
- [Background] Gami AS, Garovic VD. Contrast nephropathy after coronary angiography. Mayo Clin Proc. 2004 Feb;79(2):211-9. doi: 10.4065/79.2.211. PMID 14959916
- [Background] Goldenberg I, Shechter M, Matetzky S, Jonas M, Adam M, Pres H, Elian D, Agranat O, Schwammenthal E, Guetta V. Oral acetylcysteine as an adjunct to saline hydration for the prevention of contrast-induced nephropathy following coronary angiography. A randomized controlled trial and review of the current literature. Eur Heart J. 2004 Feb;25(3):212-8. doi: 10.1016/j.ehj.2003.11.011. PMID 14972421
- [Background] Shyu KG, Cheng JJ, Kuan P. Acetylcysteine protects against acute renal damage in patients with abnormal renal function undergoing a coronary procedure. J Am Coll Cardiol. 2002 Oct 16;40(8):1383-8. doi: 10.1016/s0735-1097(02)02308-2. PMID 12392825
- [Background] Eisenberg RL, Bank WO, Hedgock MW. Renal failure after major angiography can be avoided with hydration. AJR Am J Roentgenol. 1981 May;136(5):859-61. doi: 10.2214/ajr.136.5.859. PMID 6784516
- [Background] Kelly AM, Dwamena B, Cronin P, Bernstein SJ, Carlos RC. Meta-analysis: effectiveness of drugs for preventing contrast-induced nephropathy. Ann Intern Med. 2008 Feb 19;148(4):284-94. doi: 10.7326/0003-4819-148-4-200802190-00007. PMID 18283206
- [Background] Kay J, Chow WH, Chan TM, Lo SK, Kwok OH, Yip A, Fan K, Lee CH, Lam WF. Acetylcysteine for prevention of acute deterioration of renal function following elective coronary angiography and intervention: a randomized controlled trial. JAMA. 2003 Feb 5;289(5):553-8. doi: 10.1001/jama.289.5.553. PMID 12578487
- [Background] Briguori C, Manganelli F, Scarpato P, Elia PP, Golia B, Riviezzo G, Lepore S, Librera M, Villari B, Colombo A, Ricciardelli B. Acetylcysteine and contrast agent-associated nephrotoxicity. J Am Coll Cardiol. 2002 Jul 17;40(2):298-303. doi: 10.1016/s0735-1097(02)01958-7. PMID 12106935
- [Background] Fishbane S, Durham JH, Marzo K, Rudnick M. N-acetylcysteine in the prevention of radiocontrast-induced nephropathy. J Am Soc Nephrol. 2004 Feb;15(2):251-60. doi: 10.1097/01.asn.0000107562.68920.92. PMID 14747371
- [Background] Tepel M, van der Giet M, Schwarzfeld C, Laufer U, Liermann D, Zidek W. Prevention of radiographic-contrast-agent-induced reductions in renal function by acetylcysteine. N Engl J Med. 2000 Jul 20;343(3):180-4. doi: 10.1056/NEJM200007203430304. PMID 10900277
- [Background] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204
- [Background] Recio-Mayoral A, Chaparro M, Prado B, Cozar R, Mendez I, Banerjee D, Kaski JC, Cubero J, Cruz JM. The reno-protective effect of hydration with sodium bicarbonate plus N-acetylcysteine in patients undergoing emergency percutaneous coronary intervention: the RENO Study. J Am Coll Cardiol. 2007 Mar 27;49(12):1283-8. doi: 10.1016/j.jacc.2006.11.034. Epub 2007 Mar 12. PMID 17394959
- [Background] Briguori C, Airoldi F, D'Andrea D, Bonizzoni E, Morici N, Focaccio A, Michev I, Montorfano M, Carlino M, Cosgrave J, Ricciardelli B, Colombo A. Renal Insufficiency Following Contrast Media Administration Trial (REMEDIAL): a randomized comparison of 3 preventive strategies. Circulation. 2007 Mar 13;115(10):1211-7. doi: 10.1161/CIRCULATIONAHA.106.687152. Epub 2007 Feb 19. PMID 17309916
- [Background] McCullough PA, Wolyn R, Rocher LL, Levin RN, O'Neill WW. Acute renal failure after coronary intervention: incidence, risk factors, and relationship to mortality. Am J Med. 1997 Nov;103(5):368-75. doi: 10.1016/s0002-9343(97)00150-2. PMID 9375704
- [Background] Hoffmann U, Fischereder M, Kruger B, Drobnik W, Kramer BK. The value of N-acetylcysteine in the prevention of radiocontrast agent-induced nephropathy seems questionable. J Am Soc Nephrol. 2004 Feb;15(2):407-10. doi: 10.1097/01.asn.0000106780.14856.55. PMID 14747387
- [Background] Newman DJ, Thakkar H, Edwards RG, Wilkie M, White T, Grubb AO, Price CP. Serum cystatin C measured by automated immunoassay: a more sensitive marker of changes in GFR than serum creatinine. Kidney Int. 1995 Jan;47(1):312-8. doi: 10.1038/ki.1995.40. PMID 7731163